CLINICAL TRIAL: NCT01592786
Title: An Open-Label Study of the Safety and Tolerability of Memantine in Pediatric Patients With Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Brief Title: An Open-Label Safety Study of Memantine in Pediatric Patients With Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEM-MD-91
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Autism Spectrum Disorder (ASD); Autism; Autistic Disorder; Asperger's Disorder; Asperger's; Pediatric Autism; Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Keywords: Autism Spectrum Disorder (ASD); Autism; Autistic Disorder; Asperger's Disorder; Asperger's; Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS); Memantine; Pediatric Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine Hydrochloride (HCl) (Experimental): Once daily oral administration of open-label memantine for up to 48 weeks: 6-week dose-titration period followed by up to 42-week maintenance period.
  Interventions: Drug: Memantine Hydrochloride (HCl)

INTERVENTIONS:
Drug: Memantine Hydrochloride (HCl) — Memantine extended release 3-mg capsules; the dosages studied ranged from 3 - 15 mg/day; weight based dosing in 4 weight groups; oral administration. Dosing is once daily for up to 48 weeks.
  Other Names: Namenda

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of memantine in pediatric (6-12 years old) patients with autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS) and to identify responders for participation in a follow-up randomized withdrawal study.

DETAILED DESCRIPTION:
This 50-week multicenter and multinational clinical study is comprised of a 2-week screening period, a 6-week open-label dose-titration period followed by a variable duration maintenance period (up to 42 weeks).

Patients with at least 12 weeks of investigational product exposure who meet the protocol specified responder criterion at two consecutive visits separated by at least two weeks are eligible to transition to a randomized withdrawal study. A responder is defined as a patient who demonstrates at least a 10 point improvement (reduction in score) in the Social Responsiveness Scale (SRS) total raw score relative to the Visit 1 total raw score.

Weight based dose limits were selected in this study to ensure that exposure in terms of area under the curve (AUC) was less than the predefined limit of 2100 ng·h/mL which represents a 10-fold lower exposure than observed at the No observed adverse effect level (NOAEL) of 15 mg/kg/day in juvenile rats.

The weight-based dose limits in this study were as follows:

* Group A: ≥ 60 kg; maximum 15 mg/day
* Group B: 40-59 kg; maximum 9 mg/day
* Group C: 20-39 kg; maximum 6 mg/day
* Group D: < 20 kg; maximum 3 mg/day

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients.
2. Age of 6-12.
3. Meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) diagnostic criteria for autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
4. Have a family that is sufficiently organized and stable to guarantee adequate safety monitoring and continuous attendance to clinic visits for the duration of the study

Exclusion Criteria:

1. Have enrolled in Study MEM-MD-57A
2. Medical conditions that might interfere with the conduct of the study, confound interpretation of the study results, or endanger the patient's well-being.
3. Participation in any other clinical investigation using an experimental drug within 30 days of screening.
4. Having any primary psychiatric (Axis I) diagnosis other than autism, Asperger's Disorder, and PDD-NOS.
5. Meeting DSM-IV-TR criteria for bipolar I disorder, psychotic disorder not otherwise specified, posttraumatic stress disorder, schizophrenia, or major depressive disorder within the past 6 months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 906 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lateiner, MS, MBA, Study Director — Forest Research Institute, Inc.- A Subsidiary of Forest Laboratories, Inc.
Locations (118):
- United States (72):
  - Forest Investigative Site 068, Dothan, Alabama
  - Forest Investigative Site 005, Phoenix, Arizona
  - Forest Investigative Site 055, Tucson, Arizona
  - Forest Investigative Site 077, Little Rock, Arkansas
  - Forest Investigative Site 054, Glendale, California
  - Forest Investigative Site 109, Imperial, California
  - Forest Investigative Site 066, Irvine, California
  - Forest Investigative Site 096, Los Angeles, California
  - Forest Investigative Site 021, San Francisco, California
  - Forest Investigative Site 026, Santa Ana, California
  - Forest Investigative Site 002, Stanford, California
  - Forest Investigative Site 078, Boulder, Colorado
  - Forest Investigative Site 073, Centennial, Colorado
  - Forest Investigative Site 052, Washington D.C., District of Columbia
  - Forest Investigative Site 075, Bradenton, Florida
  - Forest Investigative Site 080, Gainesville, Florida
  - Forest Investigative Site 117, Jacksonville, Florida
  - Forest Investigative Site 065, Maitland, Florida
  - Forest Investigative Site 118, Miami, Florida
  - Forest Investigative Site 085, Oakland Park, Florida
  - Forest Investigative Site 115, Orange City, Florida
  - Forest Investigative Site 124, Orlando, Florida
  - Forest Investigative Site 125, Orlando, Florida
  - Forest Investigative Site 062, Orlando, Florida
  - Forest Investigative Site 114, Orlando, Florida
  - Forest Investigative Site 067, Tampa, Florida
  - Forest Investigative Site 101, Wellington, Florida
  - Forest Investigative Site 102, Libertyville, Illinois
  - Forest Investigative Site 023, Naperville, Illinois
  - Forest Investigative Site 082, Evansville, Indiana
  - Forest Investigative Site 123, Fort Wayne, Indiana
  - Forest Investigative Site 056, Indianapolis, Indiana
  - Forest Investigative Site 084, Indianapolis, Indiana
  - Forest Investigative Site 106, Wichita, Kansas
  - Forest Investigative Site 061, Louisville, Kentucky
  - Forest Investigative Site 074, Owensboro, Kentucky
  - Forest Investigative Site 095, Lake Charles, Louisiana
  - Forest Investigative Site 091, New Orleans, Louisiana
  - Forest Investigative Site 086, Rockville, Maryland
  - Forest Investigative Site 059, Newton, Massachusetts
  - Forest Investigative Site 108, Springfield, Massachusetts
  - Forest Investigative Site 116, Lincoln, Nebraska
  - Forest Investigative Site 097, Lincoln, Nebraska
  - Forest Investigative Site 130, Henderson, Nevada
  - Forest Investigative Site 104, Las Vegas, Nevada
  - Forest Investigative Site 136, Neptune City, New Jersey
  - Forest Investigative Site 127, Toms River, New Jersey
  - Forest Investigative Site 081, Albuquerque, New Mexico
  - Forest Investigative Site 107, Albuquerque, New Mexico
  - Forest Investigative Site 098, The Bronx, New York
  - Forest Investigative Site 072, Chapel Hill, North Carolina
  - Forest Investigative Site 069, Avon Lake, Ohio
  - Forest Investigative Site 001, Columbus, Ohio
  - Forest Investigative Site 019, Oklahoma City, Oklahoma
  - Forest Investigative Site 092, Tulsa, Oklahoma
  - Forest Investigative Site 053, Gresham, Oregon
  - Forest Investigative Site 132, Johnstown, Pennsylvania
  - Forest Investigative Site 131, McMurray, Pennsylvania
  - Forest Investigative Site 100, Media, Pennsylvania
  - Forest Investigative Site 105, Charleston, South Carolina
  - Forest Investigative Site 090, Memphis, Tennessee
  - Forest Investigative Site 057, Nashville, Tennessee
  - Forest Investigative Site 051, Houston, Texas
  - Forest Investigative Site 070, The Woodlands, Texas
  - Forest Investigative Site 028, Clinton, Utah
  - Forest Investigative Site 141, Ogden, Utah
  - Forest Investigative Site 029, Salt Lake City, Utah
  - Forest Investigative Site 064, Charlottesville, Virginia
  - Forest Investigative Site 113, Norfolk, Virginia
  - Forest Investigative Site 071, Bothell, Washington
  - Forest Investigative Site 119, Charleston, West Virginia
  - Forest Investigative Site 063, Middleton, Wisconsin
- Forest Investigative Site 177, Camperdown, New South Wales, Australia
- Belgium (4):
  - Forest Investigative Site 204, Brussels
  - Forest Investigative Site 203, Brussels
  - Forest Investigative Site 202, Hoboken
  - Forest Investigative Site 201, Leuven
- Forest Investigative Site 155, Toronto, Ontario, Canada
- Colombia (3):
  - Forest Investigative Site 227, Barranquilla
  - Forest Investigative Site 228, Bello
  - Forest Investigative Site 226, Bogotá
- Forest Investigative Site 276, Tallinn, Estonia
- France (2):
  - Forest Investigative Site 329, Bron, Rhone
  - Forest Investigative Site 326, Paris
- Hungary (6):
  - Forest Investigative Site 379, Budapest
  - Forest Investigative Site 381, Budapest
  - Forest Investigative Site 376, Budapest
  - Forest Investigative Site 378, Budapest
  - Forest Investigative Site 382, Gyula
  - Forest Investigative Site 380, Szeged
- Forest Investigative Site 401, Kopavogur, Iceland
- Italy (2):
  - Forest Investigative Site 453, Roma, Roma
  - Forest Investigative Site 452, Siena, Siena
- Forest Investigative Site 526, Wellington, New Zealand
- Poland (5):
  - Forest Investigative Site 579, Gdansk
  - Forest Investigative Site 578, Gdansk
  - Forest Investigative Site 580, Kielce
  - Forest Investigative Site 576, Kobierzyce
  - Forest Investigative Site 577, Warsaw
- Serbia (4):
  - Forest Investigative Site 626, Belgrade
  - Forest Investigative Site 627, Belgrade
  - Forest Investigative Site 629, Niš
  - Forest Investigative Site 628, Novi Sad
- Forest Investigative Site 651, Singapore, Singapore
- Forest Investigative Site 676, Cape Town, Western Cape, South Africa
- South Korea (4):
  - Forest Investigative Site 704, Yangsan, Gyeongsangnam-do
  - Forest Investigative Site 702, Seoul
  - Forest Investigative Site 703, Seoul
  - Forest Investigative Site 701, Seoul
- Spain (4):
  - Forest Investigative Site 729, Barcelona, Barcelona
  - Forest Investigative Site 728, Sabadell, Barcelona
  - Forest Investigative Site 727, Madrid, Madrid
  - Forest Investigative Site 730, Torremolinos, Málaga
- Ukraine (5):
  - Forest Investigative Site 802, Kherson, Vil. Stepanivka
  - Forest Investigative Site 803, Donetsk
  - Forest Investigative Site 807, Kharkiv
  - Forest Investigative Site 804, Kyiv
  - Forest Investigative Site 801, Odesa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over an eleven month period, from June of 2012 to May of 2013, at 118 study sites, located in the United States and 17 other countries.
Pre-assignment Details: Enrolled patients went through a 2-week screening period.
Groups:
- Memantine Hydrochloride (HCl): Memantine Hydrochloride (HCl) extended-release 3-mg capsules once daily oral administration. Dosing was 3-mg, 6-mg, 9-mg, 12-mg, or 15-mg per day, based upon patient weight.
Period: Overall Study
Arm/Group | Memantine Hydrochloride (HCl)
Started | 903 (Participants in the Safety Population are being presented.)
Completed | 765
Not Completed | 138
Not completed — Adverse Event | 60
Not completed — Lack of Efficacy | 19
Not completed — Protocol Violation | 14
Not completed — Withdrawal by Subject | 23
Not completed — Lost to Follow-up | 19
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: A total of 906 patients were enrolled in the open-label study. Of these, 903 patients received at least 1 dose of open-label treatment to comprise the Safety Population. 868 patients in the Safety Population also had at least 1 post-Visit 1 assessment of the SRS total raw score to comprise the Intent to Treat (ITT) population
Groups:
- Memantine Hydrochloride (HCl): Memantine Hydrochloride (HCl) extended-release 3-mg capsules once daily, oral administration. Dosing was 3-mg, 6-mg, 9-mg, 12-mg, or 15-mg per day, based upon patient weight.
Arm/Group | Memantine Hydrochloride (HCl)
Number analyzed (Participants) | 903
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.0 (1.9)
Sex/Gender, Customized [Number; unit: participants]
  Male | 759
  Female | 144
Race/Ethnicity, Customized [Number; unit: participants]
  White | 768
  Black or African American | 54
  Asian | 54
  American Indian or Alaska Native | 2
  Native Hawaiian or Other Pacific Islander | 3
  Other | 22
  Hispanic or Latino | 102
  Not Hispanic or Latino | 801
Region of Enrollment [Number; unit: participants]
  United States | 712
  Australia | 0
  Belgium | 11
  Canada | 1
  Colombia | 8
  Estonia | 6
  France | 14
  Hungary | 20
  Iceland | 5
  Italy | 6
  Korea, Republic of | 25
  New Zealand | 2
  Poland | 37
  Serbia | 21
  Singapore | 0
  South Africa | 2
  Spain | 17
  Ukraine | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Confirmed Social Responsiveness Scale (SRS) Responders
Description: A confirmed SRS responder was defined as a patient who had at least 12 weeks of exposure to memantine, and a ≥ 10-point reduction in the SRS total raw score relative to baseline at 2 consecutive visits separated by at least 2 weeks.
  The SRS is a 65-item, caregiver-rated assessment scale that measures observable items on social behavior and social language use, as well as characteristics of autism in a naturalistic social setting. Each item is rated on a scale from 0 (never true) to 3 (almost always true). The SRS total raw score ranges from 0 to 195; a higher score indicates greater severity of social impairment.
Time Frame: Visit 1 (Baseline) to Visit 8 (week 48/Final Visit)
Population: Of the 906 patients who enrolled in the study 903 received at least 1 dose of open-label treatment to comprise the Safety Population. The Intent to Treat (ITT) population included the 868 patients in the Safety population who also had at least 1 post-Visit 1 assessment of the SRS total raw score.
Measure: Number; unit: participants
Groups:
- Memantine Hydrochloride (HCl): Memantine Hydrochloride (HCl) extended-release 3-mg capsules once daily, oral administration. Dosing was 3-mg, 6-mg, 9-mg, 12-mg or 15-mg per day, based upon patient weight.
Arm/Group | Memantine Hydrochloride (HCl)
Number analyzed (Participants) | 868
participants
  Responders | 517
  Non responders | 351

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 14 month period from June 2012 to August 2013 at 118 study sites in the US and 17 other countries.
Groups:
- Memantine Hydrochloride (HCl): Memantine Hydrochloride (HCl) extended-release 3-mg capsules, oral administration. Dosing was 3-mg, 6-mg, 9-mg, 12-mg or 15-mg, once per day, based upon patient weight.
Arm/Group | Memantine Hydrochloride (HCl)
Serious Adverse Events (participants affected / at risk) | 6/903
Other Adverse Events (participants affected / at risk) | 196/903
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine Hydrochloride (HCl) (N=903)
Abnormal behaviour (Psychiatric disorders) | 2
Accidental exposure (Injury, poisoning and procedural complications) | 1
Constipation (Gastrointestinal disorders) | 1
Disinhibition (Psychiatric disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine Hydrochloride (HCl) (N=903)
Pyrexia (General disorders) | 52
Irritability (General disorders) | 49
Nasopharyngitis (Infections and infestations) | 57
Headache (Nervous system disorders) | 72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.